CLINICAL TRIAL: NCT04158245
Title: Changes in 18F-fluciclovine Positron Emission Tomography (PET) in Patients With Metastatic Castration Resistant Prostate Cancer Treated With With Life Prolonging Therapies: A Pilot Study
Brief Title: 18F-fluciclovine PET in Metastatic Castration Resistant Prostate Cancer Treated With Life Prolonging Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BED-IIT-382
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: Describe the changes in the 18F-fluciclovine Positron Emission Tomography (PET) in patients with metastatic castration resistant prostate cancer treated with abiraterone acetate-prednisone, enzalutamide or docetaxel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-fluciclovine PET Scan (Experimental): Single intravenous administration of 18F-fluciclovine for PET Scan.
  Interventions: Drug: 18F-fluciclovine PET Scan

INTERVENTIONS:
Drug: 18F-fluciclovine PET Scan — The use of 18F-fluciclovine PET scanning will allow a more sensitive assessment of mCRPC patients at the initiation of systemic therapy and changes observed in 18F-fluciclovine PET will correlate better with the serologic changes in PSA, allowing superior disease monitoring, as compared to conventional imaging modalities. In addition, 18F-fluciclovine PET will detect heterogeneity in disease response and thus identify potential lesions amenable to targeted therapy.
  Other Names: Axumin

SUMMARY:
This is a pilot phase 2 single-arm study, of men with metastatic castration-resistant prostate cancer (mCRPC). Patients will be treated with any of the approved life-prolonging therapies: abiraterone 1000 mg daily plus prednisone 5 mg (or dexamethasone 0.5 mg) daily, enzalutamide 160 mg daily, or docetaxel 50 mg/m2 every two weeks or 75 mg/m2 every three weeks.

DETAILED DESCRIPTION:
Prostate cancer is a hormonally-driven disease and androgens are key in the growth of both normal prostate and prostate cancer cells. Once mCRPC is evident, most patients receive a second-generation hormonal therapy to further suppress the synthesis or androgens (abiraterone) and to block androgen receptor (AR) activation, nuclear translocation and DNA binding (enzalutamide).

Conventional imaging of prostate cancer has limitations in staging, restaging after biochemical relapse, and response assessment. Functional imaging with positron emission tomography (PET) can target various aspects of tumor biology and is clearly superior in the detection of extra-prostatic disease. 18F-fluciclovine is a synthetic amino acid transported across mammalian cell membranes by amino acid transporters that are upregulated in prostate cancer cells.

18F-fluciclovine is approved for PET imaging to identify sites of prostate cancer recurrence in men with rising prostate specific antigen (PSA) following prior definitive treatment. This study describes the changes in 18F-fluciclovine PET scan and compare these results with PSA and conventional computerized tomography (CT) and bone scans, in mCRPC patients treated with abiraterone acetate-prednisone, enzalutamide or docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2;
2. Age ≥ 18 years;
3. Histologically confirmed adenocarcinoma of the prostate;
4. Ongoing use of luteinizing hormone-releasing hormone (LHRH) required in the absence of surgical castration and castrate concentration of testosterone (< 50 ng/dL);
5. Detectable PSA of at least 2 ng/dL;
6. Metastatic disease documented by CT or bone scan within 42 days of cycle 1 day 1;
7. Life expectancy of ≥ 6 months;
8. Must have disease progression despite a castrate concentration of testosterone of < 50 ng/dL based on:

   A. PSA progression defined as increase in PSA of at least 2 ng/dL and 25% from nadir values of prior therapy, determined by 2 separate measurement taken at least 1 week apart;

   And/or

   B. Radiographic disease progression based on response evaluation criteria in solid tumors (RECIST) 1.1 for soft tissue disease and/or prostate cancer working group 3 (PCWG3) for bone only disease;
9. No prior life-prolonging therapies for mCRPC are allowed, except Sipuleucel-T;
10. The use of docetaxel in the metastatic hormone-sensitive prostate cancer (mHSPC) setting is allowed;
11. Low dose prednisone (10 mg or less) or equivalent is allowed;
12. Acceptable liver function (within 28 days from enrollment) defined as:

    A. Bilirubin < 2.5 times upper limit of normal (ULN), except for patients with known Gilbert disease (in such cases bilirubin < 5 times ULN);

    B. AST (SGOT) and ALT (SGPT) < 3 times ULN
13. Acceptable renal function (within 28 days from enrollment):

    A. Serum creatinine ≤ 2.0 x ULN or creatinine clearance ≥ 30 mL/min
14. Acceptable hematologic status (within 28 days from enrollment):

    A. Absolute neutrophil count (ANC) ≥ 1000 cell/mm3 (100 x 109/L)

    B. Platelet count ≥ 100,000 platelet/mm3 (100 x 109/L)

    C. Hemoglobin ≥ 9 g/dL
15. At least 2 weeks since prior radiation before starting study treatment (cycle 1 day 1);
16. Able to understand and willing to sign a written informed consent document;
17. Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last dose of abiraterone acetate.

Exclusion Criteria:

1. Pathological findings consistent with small cell carcinoma of the prostate;
2. Prior treatment with docetaxel for metastatic castration-resistant prostate cancer (CRPC);
3. Patient with normal 18F-flucicolovine PET/CT scans at baseline;
4. Know allergies, hypersensitivity, or intolerance to abiraterone, prednisone, 18F-fluciclovine or their excipients;
5. Any chronic medical condition requiring ≥ 10 mg daily of systemic prednisone (or equivalent);
6. Major surgery (e.g., required general anesthesia) within 2 weeks before screening;
7. Uncontrolled active infection (including hepatitis B or C or AIDS). Patients with hepatitis B/C who have disease under control and no significant liver function impairment, and undetectable viral load will be allowed to participate. Similarly, patients with known HIV and ≥ 400 CD4 + T cells are allowed to participate;
8. Evidence of other metastatic malignancies within the last year;
9. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.

Ages: 18 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lewis, MD, MPH, FACP, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane Cancer Center Clinic, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-fluciclovine PET Scan: Single intravenous administration of 18F-fluciclovine for positron emission computed tomography (PET) Scan.
  18F-fluciclovine PET Scan: The use of 18F-fluciclovine PET scanning will allow a more sensitive assessment of mCRPC patients at the initiation of systemic therapy and changes observed in 18F-fluciclovine PET will correlate better with the serologic changes in prostate-specific antigen (PSA), allowing superior disease monitoring, as compared to conventional imaging modalities. In addition, 18F-fluciclovine PET will detect heterogeneity in disease response and thus identify potential lesions amenable to targeted therapy.
Period: Overall Study
Arm/Group | 18F-fluciclovine PET Scan
Started | 9
Completed | 8
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | 18F-fluciclovine PET Scan
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.56 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Haemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.23 (1.73)
Platelets [Mean (Standard Deviation); unit: cells/mcL] | 257.56 (105.58)
Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.31 (0.50)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.15 (0.56)
Alkaline phosphatase [Mean (Standard Deviation); unit: IU/L] | 95.78 (35.82)
Prostate-Specific Antigen [Mean (Standard Deviation); unit: ng/mL] | 150 (399)
Testosterone [Count of Participants; unit: Participants]
  Testosterone undetectable | 8
  Testosterone detectable | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes in 18F-fluciclovine PET Scan for Patients With mCRPC on Treatment With Life Prolonging Therapies
Description: To describe the 18F-fluciclovine PET findings for patients with mCRPC prior to starting treatment with Life Prolonging Therapies, and at 12 weeks after Life Prolonging Therapies treatment initiation. We have 4 categories that can be seen in the scan to measure the metabolic response using PERSIST 1.1, 1)stable disease, 2)progressive disease, 3)partial response and 4)complete response.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET Scan
Number analyzed (Participants) | 8
Participants
  Stable disease | 5
  Progressive disease | 0
  Partial response | 3
  Complete response | 0

2. Primary Outcome: PET Scan vs. Conventional CT and Bone Scan
Description: A comparison of 18F-fluciclovine PET with conventional CT and bone scans for patients with mCRPC prior to starting treatment with life prolonging therapies, and at 12 weeks after starting life prolonging therapies; and to correlate these changes with PSA response and progression after starting life prolonging therapies.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluciclovine PET Scan
Number analyzed (Participants) | 8
Participants
  PET scan positivity | 8
  Conventional CT scan positivity | 3
  Conventional bone scan positivity | 8
  PSA response | 3

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | 18F-fluciclovine PET Scan
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT04158245/Prot_001.pdf